CLINICAL TRIAL: NCT00700635
Title: Exploratory Evaluation of a Two-dose Schedule Versus a One-dose Schedule of Menactra® (Meningococcal [Groups A, C, Y and W 135] Polysaccharide Diphtheria Toxoid Conjugate Vaccine) in Children in the US
Brief Title: Dose Comparison Study of Menactra® in US Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA61
Record Dates: First submitted 2008-05-07; First posted 2008-06-19 (Estimated); Results first posted 2010-12-23 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Meningitis; Meningococcal Infection; Neisseria Meningitidis
Keywords: Meningitis; Meningococcal infection, Neisseria meningitidis
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Menactra® Group 1 (Experimental): Participants aged 2 to < 4 years
  Interventions: Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Conjugate
- Menactra® Group 2 (Experimental): Participants aged 4 to < 6 years
  Interventions: Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Conjugate
- Menactra® Group 3 (Active Comparator): Participants aged 6 to < 11 years
  Interventions: Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Conjugate

INTERVENTIONS:
Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Conjugate — 0.5 mL, 2 doses Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Group 1
Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Conjugate — 0.5 mL, 2 doses Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Group 2
Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Conjugate — 0.5 mL, 1 dose Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Group 3

SUMMARY:
To explore the potential benefit of the administration of Menactra vaccine as a two-dose regimen to children.

Primary Objective:

To assess, by age group, the immune response to Menactra vaccine after each vaccine injection.

DETAILED DESCRIPTION:
This is an open-label trial designed to explore the immune response to a two-dose schedule of Menactra vaccine compared with a standard one-dose schedule in children.

ELIGIBILITY:
Inclusion Criteria :

* Aged 2 to < 11 years on the day of inclusion.
* Provision of assent form signed by the subject (depending on age) and informed consent form signed by the parent(s) or another legally acceptable representative.
* Subject and parent/legal guardian able to attend all scheduled visits and comply with all trial procedures.

Exclusion Criteria :

* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine.
* Participation in the active (i.e., treatment) portion of another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy.
* Suspected or known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to a product containing any of the substances present in the study vaccine .
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator.
* Receipt of blood or blood-derived products in the past 3 months.
* Received any vaccine (other than desensitization therapy for allergies or influenza vaccine within 2 weeks before vaccination) in the 4 weeks preceding the first trial vaccination.
* Planned receipt of any vaccine within the 4 weeks following any trial vaccination(s).
* Known human immunodeficiency virus (HIV), hepatitis B surface antigen (HBs antigen), or hepatitis C seropositivity.
* History of invasive meningococcal infection (confirmed either clinically, serologically, or microbiologically).
* Thrombocytopenia, coagulation disorder, or anticoagulant use in the 3 weeks preceding inclusion contraindicating intramuscular (IM) vaccination.
* Anticipated to receive oral or injected antibiotic therapy within the 72 hours prior to any of the trial blood draws.
* Personal or family history of Guillain-Barré Syndrome (GBS).
* Any condition which, in the opinion of the Investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 333 (Actual)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (15):
- United States (15):
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Boca Raton, Florida
  - Viera, Florida
  - Woburn, Massachusetts
  - Las Vegas, Nevada
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Kingsport, Tennessee
  - Fort Worth, Texas
  - San Antonio, Texas
  - Orem, Utah
  - Midlothian, Virginia
  - Spokane, Washington

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 17 June 2008 to 25 July 2008 in 13 of 15 medical centers in the US.
Pre-assignment Details: A total of 333 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Menactra® Group 1: Participants aged 2 to less than 4 years who received 2 doses of vaccine
- Menactra® Group 2: Participants aged 4 to less than 6 years who received 2 doses of vaccine
- Menactra® Group 3: Participants aged 6 to less than 11 years who received a single dose of vaccine
Period: Overall Study
Arm/Group | Menactra® Group 1 | Menactra® Group 2 | Menactra® Group 3
Started | 111 | 111 | 111
Completed | 100 | 103 | 110
Not Completed | 11 | 8 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Protocol Violation | 2 | 2 | 0
Not completed — Withdrawal by Subject | 7 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menactra® Group 1 | Menactra® Group 2 | Menactra® Group 3 | Total
Number analyzed (Participants) | 111 | 111 | 111 | 333
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 111 | 111 | 111 | 333
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 2.46 (0.5) | 4.46 (0.5) | 8.05 (1.31) | 4.99 (2.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 55 | 53 | 158
  Male | 61 | 56 | 58 | 175
Region of Enrollment [Number; unit: participants]
  United States | 111 | 111 | 111 | 333

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Meningococcal Antibody Titers ≥ 8 After Each Vaccination
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by serum bactericidal assay using human complement (SBA-HC)
Time Frame: 30 days post-vaccination
Population: Serum bactericidal assay human complement antibody titers to each of the 4 meningococcal serogroups in the vaccine were evaluated in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Menactra® Group 1 | Menactra® Group 2 | Menactra® Group 3
Number analyzed (Participants) | 82 | 89 | 108
Percentage of Participants
  Serogroup A Post-dose 1 ≥ 8 [n = 82, 89, 107] | 59 | 36 | 65
  Serogroup A Post-dose 2 ≥ 8 [n = 81, 89, 0] | 83 | 67 | NA — Dose 2 vaccination was not administered to the Menactra Group 3
  Serogroup C Post-dose 1 ≥ 8 [n = 82, 89, 108] | 72 | 51 | 62
  Serogroup C Post-dose 2 ≥ 8 [n = 82, 89, 0] | 95 | 88 | NA — Dose 2 vaccination was not administered to the Menactra Group 3
  Serogroup Y Post-dose 1 ≥ 8 [n = 82, 89, 108] | 60 | 65 | 71
  Serogroup Y Post-dose 2 ≥ 8 [n = 82, 89, 0] | 100 | 96 | NA — Dose 2 vaccination was not administered to the Menactra Group 3
  Serogroup W-135 Post-dose 1 ≥ 8 [n = 82, 89, 108] | 66 | 79 | 91
  Serogroup W-135 Post-dose 2 ≥ 8 [n = 82, 89, 0] | 96 | 96 | NA — Dose 2 vaccination was not administered to the Menactra Group 3

2. Secondary Outcome: Percentage of Participants With Meningococcal Antibody Titers at ≥ 4 After Each Vaccination
Description: as for outcome 1
Time Frame: 30 days post-vaccination
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Menactra® Group 1 | Menactra® Group 2 | Menactra® Group 3
Number analyzed (Participants) | 82 | 89 | 108
Percentage of Participants
  Serogroup A Post-dose 1 ≥ 4 [n = 82, 89, 107] | 73 | 58 | 79
  Serogroup A Post-dose 2 ≥ 4 [n = 81, 89, 0] | 94 | 79 | NA — Dose 2 vaccination was not administered to the Menactra Group 3
  Serogroup C Post-dose 1 ≥ 4 [n = 82, 89, 108] | 78 | 63 | 69
  Serogroup C Post-dose 2 ≥ 4 [n = 82, 89, 0] | 95 | 91 | NA — Dose 2 vaccination was not administered to the Menactra Group 3
  Serogroup Y Post-dose 1 ≥ 4 [n = 82, 89, 108] | 77 | 83 | 83
  Serogroup Y Post-dose 2 ≥ 4 [n = 82, 89, 0] | 100 | 98 | NA — Dose 2 vaccination was not administered to the Menactra Group 3
  Serogroup W-135 Post-dose 1 ≥ 4 [n = 82, 89, 108] | 83 | 89 | 96
  Serogroup W-135 Post-dose 2 ≥ 4 [n = 82, 89, 0] | 99 | 100 | NA — Dose 2 vaccination was not administered to the Menactra Group 3

3. Secondary Outcome: Geometric Mean Titers (GMTs) of Meningococcal Antibodies After Each Menactra® Vaccination.
Description: as for outcome 1
Time Frame: 30 days post-vaccination
Population: Geometric mean titers (GMTs) of Serum Bactericidal Assay Human Complement (SBA-HC) for the vaccine Serogroups were analyzed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menactra® Group 1 | Menactra® Group 2 | Menactra® Group 3
Number analyzed (Participants) | 82 | 89 | 108
Titers
  Serogroup A Post-dose 1 [n = 82, 89, 107] | 9.97 [7.37 to 13.5] | 5.59 [4.35 to 7.18] | 12.7 [9.53 to 16.8]
  Serogroup A Post-dose 2 [n = 81, 89, 0] | 24.3 [17.4 to 33.9] | 13.6 [9.77 to 18.9] | NA [NA to NA] — Dose 2 vaccination was not administered to the Menactra Group 3.
  Serogroup C Post-dose 1 [n = 82, 89, 108] | 13.4 [9.76 to 18.4] | 8.99 [6.41 to 12.6] | 18.5 [12.1 to 28.4]
  Serogroup C Post-dose 2 [n = 82, 89, 0] | 92.8 [65.5 to 132] | 46.1 [32.7 to 65.2] | NA [NA to NA] — Dose 2 vaccination was not administered to the Menactra Group 3.
  Serogroup Y Post-dose 1 [n = 82, 89, 108] | 8.42 [6.51 to 10.9] | 9.13 [7.27 to 11.5] | 14.2 [10.8 to 18.6]
  Serogroup Y Post-dose 2 [n = 82, 89, 0] | 78.4 [62.4 to 98.6] | 42.0 [32.1 to 55.0] | NA [NA to NA] — Dose 2 vaccination was not administered to the Menactra Group 3.
  Serogroup W-135 Post-dose 1 [n = 82, 89, 108] | 12.4 [9.33 to 16.5] | 15.5 [11.9 to 20.2] | 24.1 [19.1 to 30.5]
  Serogroup W-135 Post-dose 2 [n = 82, 89, 0] | 57.8 [44.2 to 75.7] | 50.3 [37.9 to 66.8] | NA [NA to NA] — Dose 2 vaccination was not administered to the Menactra Group 3.

4. Secondary Outcome: Percentage of Participants Reporting Solicited Injection Site and Solicited Systemic Reactions After Dose 1 Vaccination
Description: Solicited injection site reactions: Erythema, Swelling, Pain. Solicited systemic reactions: Fever (temperature), Headache, Malaise, and Myalgia.
Time Frame: 7 days post-vaccination 1
Population: Safety analysis was on all enrolled and vaccinated participants, intent-to-treat population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Menactra® Group 1 | Menactra® Group 2 | Menactra® Group 3
Number analyzed (Participants) | 111 | 111 | 111
Percentage of Participants
  Any Solicited Injection Site Reaction Post Dose 1 | 67 | 60 | 67
  Any Pain | 53 | 53 | 58
  Grade 3 Pain (Incapacitating) | 1 | 0 | 2
  Any Erythema | 47 | 27 | 32
  Grade 3 Erythema (≥ 5 cm) | 5 | 4 | 8
  Any Swelling | 23 | 18 | 23
  Grade 3 Swelling (≥ 5 cm) | 4 | 3 | 5
  Any Solicited Systemic Reaction Post Dose 1 | 52 | 43 | 38
  Any Fever | 7 | 4 | 1
  Grade 3 Fever (> 39.0 ºC or > 102.2 ºF) | 1 | 1 | 0
  Any Headache | 7 | 15 | 23
  Grade 3 Headache (Prevents daily activities) | 0 | 0 | 0
  Any Vomiting | 6 | 4 | 2
  Grade 3 Vomiting (≥ 3 episodes per 24 hours) | 0 | 1 | 0
  Any Drowsiness | 21 | 16 | 14
  Grade 3 Drowsiness (Disabling) | 1 | 4 | 0
  Any Anorexia | 20 | 10 | 7
  Grade 3 Anorexia (Skips ≥ 3 meals) | 0 | 0 | 0
  Any Irritability | 35 | 20 | 11
  Grade 3 Irritability (>3 hours duration) | 2 | 4 | 2
  Any Arthralgia | 7 | 8 | 7
  Grade 3 Arthralgia (Unwllling to move due to pain) | 0 | 0 | 1
  Any Diarrhea | 17 | 8 | 3
  Grade 3 Diarrhea (≥ 5 episodes per 24 hours) | 2 | 0 | 0

5. Secondary Outcome: Percentage of Participants Reporting Solicited Injection Site and Solicited Systemic Reactions After Dose 2 Vaccination
Description: as for outcome 4
Time Frame: 7 days post-vaccination 2
Population: Safety analysis was on all enrolled and vaccinated participants, intent-to-treat population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Menactra® Group 1 | Menactra® Group 2 | Menactra® Group 3
Number analyzed (Participants) | 111 | 111 | 0
Percentage of Participants
  Any Solicited Injection Site Reaction Post Dose 2 | 60 | 64 |
  Any Pain | 48 | 52 |
  Grade 3 Pain (Incapacitating) | 0 | 1 |
  Any Erythema | 37 | 36 |
  Grade 3 Erythema (≥ 5 cm) | 8 | 4 |
  Any Swelling | 20 | 15 |
  Grade 3 Swelling (≥ 5 cm) | 3 | 2 |
  Any Solicited Systemic Reaction Post Dose 2 | 53 | 49 |
  Any Fever | 5 | 13 |
  Grade 3 Fever (> 39.0 ºC or > 102.2 ºF) | 0 | 3 |
  Any Headache | 6 | 14 |
  Grade 3 Headache (Prevents daily activities) | 0 | 1 |
  Any Vomiting | 5 | 7 |
  Grade 3 Vomiting (≥ 3 episodes per 24 hours) | 1 | 2 |
  Any Drowsiness | 19 | 18 |
  Grade 3 Drowsiness (Disabling) | 1 | 2 |
  Any Anorexia | 21 | 17 |
  Grade 3 Anorexia (Skips ≥ 3 meals) | 1 | 1 |
  Any Irritability | 31 | 23 |
  Grade 3 Irritability (>3 hours duration) | 5 | 3 |
  Any Arthralgia | 8 | 7 |
  Grade 3 Arthralgia (Unwllling to move due to pain) | 0 | 0 |
  Any Diarrhea | 15 | 7 |
  Grade 3 Diarrhea (≥ 5 episodes per 24 hours) | 0 | 0 |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the day of vaccination (Day 0) up to 6 months post-dose 2 vaccination
Arm/Group | Menactra® Group 1 | Menactra® Group 2 | Menactra® Group 3
Serious Adverse Events (participants affected / at risk) | 4/111 | 3/111 | 0/111
Other Adverse Events (participants affected / at risk) | 58/111 | 57/111 | 64/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menactra® Group 1 (N=111) | Menactra® Group 2 (N=111) | Menactra® Group 3 (N=111)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Breath holding (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Menactra® Group 1 (N=111) | Menactra® Group 2 (N=111) | Menactra® Group 3 (N=111)
Diarrhea (Gastrointestinal disorders) | 19/109 (19) | 9/108 (9) | 3 (3)
Vomiting (Gastrointestinal disorders) | 6/109 (6) | 7/103 (7) | 2 (2)
Injection site erythma (General disorders) | 51/109 (51) | 37/103 (37) | 35 (35)
Fever (General disorders) | 8/109 (8) | 13/103 (13) | 1 (1)
Irritability (General disorders) | 38/109 (38) | 24/103 (24) | 12 (12)
Injection site pain (General disorders) | 58/109 (58) | 57/108 (57) | 64 (64)
Pyrexia (General disorders) | 14 (14) | 8 (8) | 3 (3)
Injection site swelling (General disorders) | 25/109 (25) | 19/108 (19) | 25 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8/109 (8) | 9/108 (9) | 8 (8)
Drowsiness (Nervous system disorders) | 23/109 (23) | 18/103 (18) | 16 (16)
Headache (Nervous system disorders) | 8/109 (8) | 16/108 (16) | 25 (25)
Anorexia (Psychiatric disorders) | 22/109 (22) | 17/103 (17) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (25) | 15 (16) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 4 (4) | 0 (0)
Injection site induration (General disorders) | 7 (7) | 5 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (7) | 4 (4) | 2 (2)
Otitis media (Infections and infestations) | 6 (6) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 4 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (9) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications